CLINICAL TRIAL: NCT04917939
Title: Gene Expression Changes of Brain Tissue in Human Temporal Lobe Epilepsy With Hippocampal Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0291
Record Dates: First submitted 2021-06-07; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Epilepsy; Hippocampal Sclerosis
Keywords: Epilepsy; Hippocampal Sclerosis
MeSH Terms: conditions — Epilepsy; Hippocampal Sclerosis | interventions — Sequence Analysis, RNA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- epilepsy with HS
  Interventions: Other: RNA sequencing
- epilepsy without HS
  Interventions: Other: RNA sequencing

INTERVENTIONS:
Other: RNA sequencing — Samples in both groups will be sequenced by single-cell sequencing and spatial transcription sequencing.

SUMMARY:
Epilepsy is a common neurological disease, manifested in the sudden abnormal discharge of neurons leading to short-term brain dysfunction, has become the neurology after headache the second most common disease. In China, the prevalence of epilepsy is about 4.7-8.5 per 1,000, and more than 400,000 new cases of epilepsy are developed each year. Of these, 30% of patients were treated with ineffective medication, developing into a drug-incurable epilepsy that required surgery and other treatments. The most common type of epilepsy is temporal lobe epilepsy, while the common complication in temporal lobe epilepsy is hippocampal sclerosis, which often requires surgical removal. The incidence of inner temporal lobe epilepsy associated with hippocampal sclerosis is increasing, but its exact cause and specific pathogenesis are still unclear, so clarifying its pathogenesis will contribute to the understanding of temporal lobe epilepsy and the improvement of surgical procedures. This study is intended to get single-cell transcriptome as well as spatial transcriptome data of temporal lobe and hippocampus samples. By studying gene expression change associated with epilepsy and hippocampus sclerosis, we intended to find possible prognostic-related molecules and to deepen understanding of pathological changes in epilepsy at the molecular level.

ELIGIBILITY:
Inclusion Criteria:

* Patients confirmed in our hospital as having temporal lobe epilepsy and intending surgery to remove temporal lobe and hippocampal tissue;
* Volunteer to participate in this clinical trial, comply with the requirements of this clinical trial and sign an informed consent form.

Exclusion Criteria:

* Chronic diseases of the central nervous system other than temporal lobe epilepsy;
* Other patients that are not suitable for this clinical trial determined by the researchers;

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Epilepsy patients with or without hippocampal sclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
RNA sequencing data | up to 24 weeks
  Single-cell sequencing and spatial transcription sequencing data of samples.

CONTACTS AND LOCATIONS:
Overall Officials: 2nd Affiliated Hospital, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2ndAffiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China